CLINICAL TRIAL: NCT01696513
Title: Pilot Split Face Randomized, Evaluator Blinded Study on the Effect of Subcision and Suctioning With a Microdermabrasion Device on Rolling Acne Scars
Brief Title: Effect of Subcision and Suction on Acne Scars
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, Professor in Dermatology, Otolaryngology- Head and Neck Surgery, and Surgery-Organ Transplantation, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU66710
Record Dates: First submitted 2012-09-14; First posted 2012-10-01 (Estimated); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Acne Scars
MeSH Terms: interventions — Suction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subcision & Suction (Experimental): Standard treatment for acne scars followed by suction.
  Interventions: Procedure: Suction; Procedure: Subcision
- Subcision (Active Comparator): Standard treatment for acne scars only
  Interventions: Procedure: Subcision

INTERVENTIONS:
Procedure: Suction
  Arms: Subcision & Suction
Procedure: Subcision

SUMMARY:
The primary objective of this study is to determine whether the use of standard treatment in conjunction with suction will improve acne scars compared to a standard treatment alone.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and over
* Have bilateral rolling acne scars
* Are in good health
* Subject has the willingness and ability to understand and provide informed consent for the use of their tissue and communicate with the investigator.

Exclusion Criteria:

* Under 18 years of age
* Pregnancy or lactation
* Unable to understand the protocol or give informed consent
* Has mental illness
* Recent Accutane use in the past 6 months
* Prone to hypertrophic and keloidal scarring

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-09; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in acne scarring compared to baseline after treatments | Baseline and 4 months
  The change in acne scarring is measured using a global scarring grading system to compare baseline scarring to the treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Department of Dermatology, Chicago, Illinois, United States

REFERENCES:
- [Derived] Shi VJ, Ma MS, Koza E, Haq M, Ahmed A, Yi MD, Dirr MA, Anvery N, Christensen RE, Pagdhal K, Geisler A, Nodzenski M, Roongpisuthipong W, Brieva JC, Cahn BA, Yoo SS, Lucas J, Poon E, West DP, Fife D, Alam M. Subcision with and without suction for acne scars: a split-faced, rater-blinded randomized control trial. Arch Dermatol Res. 2024 Jun 7;316(7):344. doi: 10.1007/s00403-024-03128-4. PMID 38847979